CLINICAL TRIAL: NCT00462605
Title: A Phase II Study of and Oral Histone Deacytylase Inhibitor, MS-275 (NSC 706995), in Combination With Sargramostim (GM-CSF, Berlex, Inc.) Treating Relapsed and Refractory Myeloid Malignancies
Brief Title: MS-275 and GM-CSF in Treating Patients With Myelodysplastic Syndrome and/or Relapsed or Refractory Acute Myeloid Leukemia or Acute Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00195; J06114; U01CA070095 (NIH); NCT00466115 (obsolete NCT alias)
Record Dates: First submitted 2007-04-18; First posted 2007-04-19 (Estimated); Results first posted 2017-04-17 (Actual); Last update posted 2017-07-18 (Actual); Status verified 2017-06

CONDITIONS: Adult Acute Lymphoblastic Leukemia in Remission; Adult Acute Megakaryoblastic Leukemia (M7); Adult Acute Minimally Differentiated Myeloid Leukemia (M0); Adult Acute Monoblastic Leukemia (M5a); Adult Acute Monocytic Leukemia (M5b); Adult Acute Myeloblastic Leukemia With Maturation (M2); Adult Acute Myeloblastic Leukemia Without Maturation (M1); Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Adult Acute Myelomonocytic Leukemia (M4); Adult Erythroleukemia (M6a); Adult Pure Erythroid Leukemia (M6b); Chronic Myelomonocytic Leukemia; de Novo Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasm, Unclassifiable; Previously Treated Myelodysplastic Syndromes; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Acute Myeloid Leukemia; Refractory Anemia; Refractory Anemia With Excess Blasts; Refractory Anemia With Ringed Sideroblasts; Refractory Cytopenia With Multilineage Dysplasia; Secondary Acute Myeloid Leukemia; Secondary Myelodysplastic Syndromes; Untreated Adult Acute Lymphoblastic Leukemia; Untreated Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myeloid, Acute; Congenital Abnormalities; Leukemia, Myelomonocytic, Acute; Leukemia, Erythroblastic, Acute; Leukemia, Myelomonocytic, Chronic; Myeloproliferative Disorders; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Anemia, Refractory; Anemia, Refractory, with Excess of Blasts | interventions — entinostat; sargramostim; Granulocyte-Macrophage Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): Patients receive oral MS-275 on days 1, 8, 15, and 22. Patients also receive sargramostim (GM-CSF) subcutaneously once daily on days 1-42 in courses 3 and 5 and on days 1-35 in courses 1, 2, 4, and 6. Treatment repeats every 6 weeks for 2-6 courses in the absence of disease progression or unacceptable toxicity. After completion of 2 courses of study therapy, patients who achieve a complete or partial response may receive an additional 4 courses. Patients who maintain stable disease for more than 2 months after completion of 6 courses of study therapy may receive an additional 6 courses at the time of disease progression, provided they meet original eligibility criteria.
  Interventions: Drug: entinostat; Drug: sargramostim

INTERVENTIONS:
Drug: entinostat — Given PO
  Other Names: HDAC inhibitor SNDX-275; SNDX-275
Drug: sargramostim — Given SC
  Other Names: GM-CSF; Leukine; Prokine

SUMMARY:
This phase II trial is studying how well giving MS-275 together with GM-CSF works in treating patients with myelodysplastic syndrome and/or relapsed or refractory acute myeloid leukemia. MS-275 may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the cancer. Colony-stimulating factors, such as GM-CSF, may increase the number of immune cells found in bone marrow or peripheral blood. Giving MS-275 together with GM-CSF may be an effective treatment for myelodysplastic syndrome and acute myeloid leukemia

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine clinical response in patients with myelodysplastic syndromes and/or relapsed or refractory acute myeloid leukemia or acute lymphocytic leukemia treated with MS-275 in combination with sargramostim (GM-CSF).

SECONDARY OBJECTIVES:

I. Determine the clinical activity of this regimen, in terms of changes in peripheral blood counts and changes in individual patient transfusion requirements, in these patients.

II. Determine the biologic activity of this regimen, in terms of changes in the peripheral blood and bone marrow phenotype (i.e., induction of markers of myeloid differentiation or lymphoid differentiation) and changes in detectable cytogenetic abnormalities in the blood and marrow compartments, in these patients.

III. Determine the toxicity profile of this regimen in these patients.

OUTLINE:

Patients receive oral MS-275 on days 1, 8, 15, and 22. Patients also receive sargramostim (GM-CSF) subcutaneously once daily on days 1-42 in courses 3 and 5 and on days 1-35 in courses 1, 2, 4, and 6. Treatment repeats every 6 weeks for 2-6 courses in the absence of disease progression or unacceptable toxicity.

After completion of 2 courses of study therapy, patients who achieve a complete or partial response may receive an additional 4 courses. Patients who maintain stable disease for more than 2 months after completion of 6 courses of study therapy may receive an additional 6 courses at the time of disease progression, provided they meet original eligibility criteria.

Patients undergo blood and bone marrow (BM) collection at baseline and periodically during study for biologic correlative studies. Peripheral blood and bone marrow samples are assessed for changes in progenitor phenotype and clonogenic growth by flow cytometry and for changes in cytogenetics (i.e., malignant:nonmalignant cell ratio in BM CD34-positive cells, peripheral blood monocytes, peripheral blood neutrophils, and bone marrow and peripheral blood lymphoblasts) by FISH. Terminal differentiation of CD34-positive progenitor cells is studied in vitro in long-term cultures.

After completion of study therapy, patients are followed periodically for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of 1 of the following diseases by bone marrow aspiration and/or biopsy:

  * Myelodysplastic syndromes (MDS) meeting the following criteria:
  * Must have 1 of the following subtypes:
  * Refractory anemia (RA) (no RA with 5q-syndrome),
  * RA with ringed sideroblasts or
  * Refractory cytopenia with multilineage dysplasia
* Myelodysplastic syndromes (MDS) meeting the following criteria:

Must have 1 of the following subtypes:

* Refractory cytopenia with multilineage dysplasia and ringed sideroblasts,
* RA with excess blasts (RAEB)-1, RAEB-2,
* Myelodysplastic syndromes, unclassified or
* Chronic myelomonocytic leukemia

  * International Prognostic Scoring System score of intermediate-2 or high-risk
  * Acute myeloid leukemia (AML) meeting 1 of the following criteria:
  * Relapsed or refractory AML, including any of the following subtypes:
  * * AML with recurrent cytogenetic abnormalities (i.e., AML with 11q23 [MLL] abnormalities)
* AML with multilineage dysplasia
* AML that is therapy-related
* AML, not otherwise categorized (M0 [minimally differentiated], M1 [without maturation], M2 [with maturation], M4 [myelomonocytic leukemia], M5 [monoblastic/monocytic leukemia], M6 [erythroid leukemia], and M7 [megakaryoblastic leukemia])

  * Untreated AML
* Newly diagnosed patients are eligible provided they do not qualify for potentially curative intensive chemotherapeutic regimens

  * Acute lymphocytic leukemia (ALL) meeting 1 of the following criteria:
* Relapsed or refractory ALL
* Patients with any measurable residual disease are eligible, including cytogenetic abnormalities

  * Untreated ALL
* Newly diagnosed patients are eligible provided they do not qualify for potentially curative intensive chemotherapeutic regimens, including any of the following:
* Patients who have refused chemotherapy for untreated ALL
* Patients who are deemed to be poor candidates medically for ALL induction chemotherapy

  * Relatively stable bone marrow function for > 7 days prior to study entry
* WBC count that has not doubled within the past 7 days
* WBC =<10,000/mm³

  * No uncontrolled peripheral leukemia (i.e., blast count > 30,000/mm³)
  * No active CNS disease
* Lumbar puncture with negative cytology required for patients with clinical symptoms of active CNS disease

  * Not a candidate for a potentially curative allogeneic stem cell transplantation OR considered a poor candidate for such a procedure due to age, medical comorbidities, or lack of a suitable donor
  * Hemoglobin >= 8 g/dL (transfusions allowed)
  * Creatinine =< 2.0 mg/dL
  * Bilirubin =< 1.6 mg/dL (unless secondary to hemolysis)
  * AST or ALT =< 3 times upper limit of normal (unless disease-related)
  * Not pregnant or nursing
  * Negative pregnancy test
  * Fertile patients must use effective contraception
  * No untreated or progressive infections
  * No history of intolerance to sargramostim (GM-CSF)
  * Recovered from all treatment-related toxicities
  * More than 2 weeks since prior therapy for AML, ALL, or MDS, including chemotherapy, hematopoietic growth factors, or biologic therapy such as monoclonal antibodies
  * Concurrent hydroxyurea allowed during course 1 for control of leukocytosis if WBC > 30,000/mm³
  * ECOG performance status 0-2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-04; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: B. Smith, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I
Started | 24
Completed | 10
Not Completed | 14

BASELINE CHARACTERISTICS:
Arm/Group | Arm I
Number analyzed (Participants) | 24
Age, Continuous [Median (Full Range); unit: years] | 71 [52 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 15
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Response (Complete and Partial Response) in Patients With Myeloid Disorders
Description: Response to treatment was assessed after two cycles, according to International Working Group (IWG) criteria. Cytogenetic responses were monitored in patients with abnormalities at baseline.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I
Number analyzed (Participants) | 10
Participants
  Complete Remission (CR) | 0
  Partial Remission (PR) | 1
  Hematologic Improvement in Neutrophils (HI-N) | 2
  Stable Disease (SD) | 5
  Progressive Disease (PD) | 2

2. Secondary Outcome: Clinical Activity Assessed by Change in Peripheral Blood Counts
Time Frame: Baseline and after 2 cycles
Measure: Mean (Standard Error); unit: cell/mm^3
Arm/Group | Arm I
Number analyzed (Participants) | 10
cell/mm^3
  ANC +/- SEM at baseline | 578 (126)
  ANC +/- SEM after 2 cycles | 1137 (384)

3. Secondary Outcome: Clinical Activity Assessed by Change in Transfusion Requirements
Time Frame: Baseline and after 2 cycles
Population: Due to the limited number of clinical responders, this outcome was not measured.
Arm/Group | Arm I
Number analyzed (Participants) | 0

4. Secondary Outcome: Changes in Detectable Chromosomal Abnormalities Measured by Fluorescent in Situ Hybridization (FISH)
Time Frame: Baseline and 6, 12, 24, and 36 weeks
Population: Due to the limited number of clinical responders, the research assay was not done.
Arm/Group | Arm I
Number analyzed (Participants) | 0

5. Secondary Outcome: Change in the Percentage of Cells With Normal and Abnormal Myeloid Phenotype Measured by Flow Cytometry
Time Frame: Baseline and 6, 12, 24, and 36 weeks
Population: Due to the limited number of clinical responders, the research assay was not done.
Arm/Group | Arm I
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Arm I
Serious Adverse Events (participants affected / at risk) | 19/24
Other Adverse Events (participants affected / at risk) | 6/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (N=24)
Neutropenic infection (Infections and infestations) | 5
Bone Pain (Musculoskeletal and connective tissue disorders) | 3
Fatigue (General disorders) | 2
Pericardial effusion (Cardiac disorders) | 1
Weakness (Musculoskeletal and connective tissue disorders) | 1
anorexia (Gastrointestinal disorders) | 1
hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
vasovagal episode (Nervous system disorders) | 1
Joint pain (Musculoskeletal and connective tissue disorders) | 1
cough (Respiratory, thoracic and mediastinal disorders) | 1
pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (N=24)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 2
hyponatremia (Metabolism and nutrition disorders) | 2
confusion (Nervous system disorders) | 2
Neutropenic infection (Infections and infestations) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
fatigue (General disorders) | 1
back pain (Musculoskeletal and connective tissue disorders) | 1
hypocalcemia (Metabolism and nutrition disorders) | 1
GI bleed (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less